CLINICAL TRIAL: NCT01996345
Title: Vaginal Pessary Versus Expectant Management for the Prevention of Delivery Prior to 36 Weeks in Women With Placenta Previa
Brief Title: Vaginal Pessary Versus Expectant Management for Placenta Previa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated early do to a business decision by sponsor and lack of ability to recruit the needed number of participants.
Sponsor: Pediatrix (Other)
Collaborators: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBX0028
Record Dates: First submitted 2013-11-14; First posted 2013-11-27 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Placenta Previa
Keywords: Placenta Previa; Vaginal Pessary; Premature Birth
MeSH Terms: conditions — Placenta Previa; Premature Birth

STUDY DESIGN:
Masking Description: There is no masking in this study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical Pessary Placement (Experimental): For the patients assigned to receive a cervical pessary, they will be evaluated and fitted for a pessary by the physician within 3-4 days unless exclusion criteria develop. After it is placed she will be evaluated for comfort. She will be asked to leave it in at all times but informed that removal and withdrawal from the study is always her option.
  Interventions: Procedure: Cervical Pessary Placement
- Expectant Managment (No Intervention): Each participant will have standard care for placenta previa. This is the same care that a patient with a placenta previa would ordinarily receive even if she were not participating in the trial. The trial's participating investigators agree that the management outlined in this section is standard management for placenta previa.

INTERVENTIONS:
Procedure: Cervical Pessary Placement — For the patients assigned to receive a cervical pessary, they will be evaluated and fitted for a pessary by the physician within 3-4 days unless exclusion criteria develop. After it is placed she will be evaluated for comfort. She will be asked to leave it in at all times but informed that removal and withdrawal from the study is always her option.
  Arms: Cervical Pessary Placement

SUMMARY:
The purpose of this study is to perform a large multi-center randomized trial comparing the role of vaginal pessary versus expectant management in women with placenta previa between 22w0d and 32w0d of gestation in prolonging gestation until ≥36 weeks. Secondary outcomes will assess duration of antepartum admission, total blood loss, gestational age at delivery, type of cesarean delivery, and a composite neonatal outcome. The hypothesis is that the use of a vaginal pessary in patients presenting with placenta previa between 22-32 weeks will decrease delivery prior to 36 weeks as compared to expectantly managing these patients.

DETAILED DESCRIPTION:
While the use of pessary in this scenario has not been previously assessed, it is reasonable to infer, from the data for use of pessary to prevent preterm birth, and the data regarding the efficacy of cervical cerclage in reducing bleeding and preterm birth in patients with placenta previa to this clinical conundrum. If cerclage improves pregnancy outcomes in patients with placenta previa, the use of a vaginal pessary should be a less-invasive but similarly efficacious alternative to maintain cervical length. The purpose of this study is to compare two treatment options reasonably used in clinical practice. Use of cervical pessary is not expected to increase antenatal costs beyond the minimal cost of the pessary. Additionally, given the results of the available clinical trials on cerclage maintaining cervical length and decreasing bleeding, this procedure has the potential to decrease the cost of both antepartum admissions for bleeding and neonatal care.

A substantial number of women with placenta previa will not hemorrhage until they reach the third trimester, thus, by allowing for enrollment and pessary placement as late as 32w0d, the intervention may be applied to the broadest "at risk" population. As previously mentioned literature on the use of cerclage in patients with placenta previa and short cervix are limited by a reduced number of eligible subjects and concern over safety issues has not been assuaged by these small studies. As pessary placement appears to carry little if any risk based on a number of published studies, eligibility can be expanded to any cervical length.

ELIGIBILITY:
Inclusion Criteria:

* Participant age 18 years or older
* Gestational age between 22w0d and 32w0d, inclusive, at time of enrollment
* Singleton pregnancy
* Complete Placenta Previa
* Intact Membranes
* No allergies to material in pessary
* Plan to deliver at PI's hospital
* Informed consent obtained, signed/dated

Exclusion Criteria:

* Active preterm labor
* Nonreassuring fetal heart rate tracing
* Intrauterine fetal death
* Active bleeding (may be enrolled if hemostatic >48 hours)
* Ruptured membranes
* Any fetal condition likely to cause serious neonatal morbidity independent of gestational age: Fetal malformation likely to require surgery, Fetal malformation involving vital organs, Fetal viral infection, Hydrops fetalis,
* Known Uterine Anomaly
* Cervical Cerclage present at time of enrollment
* Maternal condition that warrant continued hospitalization (example severe preeclampsia, Diabetes out of control, maternal heart disease)

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Decrease Delivery Prior to 36 weeks in patients with a gestational age of 22.0- 32.0 presenting with placenta previa. | day of birth
  This outcome, a decrease in the number of delivery that occur before 36 weeks of pregnancy who have a diagnosed placenta previa. The gestational age is noted at the time of birth.

SECONDARY OUTCOMES:
Need for packed red blood cells or hematologic product replacement | from birth to 60 days
  note the number of blood transfusions the baby received from birth until 60 days post birth
Neonate or Fetal Death | From time of trial entry to 60 days post birth (approximately 34 weeks)
  death of fetus or newborn up to 60 days post delivery
Neonatal Outcomes | From Birth to 60 days of Age
  Including birthweight, neonatal death, composite neonatal morbidity (any of the following: respiratory distress syndrome, bronchopulmonary dysplasia, severe intraventricular hemorrhage, periventricular leukomalacia, proven sepsis, necrotizing enterocolitis, or perinatal death.) and specific neonatal morbidities including: Apgar <3 at 5 min, ICU admission, , cord pH, 7.1.
Any adverse reactions to the cervical pessary. | from 0 to as many as 18 weeks.
  unexpected adverse reaction such as cervical trauma, infection, allergy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Garite, MD, Principal Investigator — Obstetrix Medical Group; Irene Stafford, MD, Principal Investigator — Baylor College of Medicine
Locations (10):
- United States (10):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Norton Kosair Children's Hospital, Louisville, Kentucky
  - Tulane - Lakeside Hospital for Women and Children, Metairie, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Baylor/Texas Children's Hospital & Pavilion, Houston, Texas
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsors Website — http://pediatrix.com